CLINICAL TRIAL: NCT06839105
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AWT020 Alone and in Combination With Other Antitumor Therapies in Patients With Advanced Malignancies
Brief Title: A Clinical Study to Evaluate the Safety and Tolerability of AWT020 in Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AWT020-001-I
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer, Colorectal Cancer, Renal Cell Carcinoma, Melanoma and Other Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Renal Cell; Melanoma | interventions — Paclitaxel; Cisplatin; Carboplatin; Pemetrexed; Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AWT020 (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: AWT020
- AWT020 combination with taxol and cisplatin or carboplatin (Experimental)
  Interventions: Drug: Taxol; Drug: Cisplatin or Carboplatin; Drug: AWT020
- AWT020 combination with Pemetrexed and cisplatin or carboplatin (Experimental)
  Interventions: Drug: Cisplatin or Carboplatin; Drug: Pemetrexed; Drug: AWT020
- AWT020 combination with Oxaliplatin,Capecitabine and Bevacizumab (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab; Drug: AWT020
- AWT020 combination with Renvastinib (Experimental)
  Interventions: Drug: Renvastinib; Drug: AWT020

INTERVENTIONS:
Drug: Taxol — 135~175 mg/m2, Q3W
  Arms: AWT020 combination with taxol and cisplatin or carboplatin
Drug: Cisplatin or Carboplatin — Cisplatin(75 mg/m2, Q3W) or Carboplatin (AUC=5~6, Q3W)
  Arms: AWT020 combination with Pemetrexed and cisplatin or carboplatin; AWT020 combination with taxol and cisplatin or carboplatin
Drug: Pemetrexed — 500 mg/m2, Q3W
  Arms: AWT020 combination with Pemetrexed and cisplatin or carboplatin
Drug: Oxaliplatin — 130 mg/m2, Q3W
  Arms: AWT020 combination with Oxaliplatin,Capecitabine and Bevacizumab
Drug: Capecitabine — 1000 mg/m2, BID, day1-14, oral, q3w
  Arms: AWT020 combination with Oxaliplatin,Capecitabine and Bevacizumab
Drug: Bevacizumab — 7.5 mg/kg, Q3W
  Arms: AWT020 combination with Oxaliplatin,Capecitabine and Bevacizumab
Drug: Renvastinib — 8mg or 20mg, QD
  Arms: AWT020 combination with Renvastinib
Drug: AWT020 — q3w or q2w, i.v.

SUMMARY:
The purpose of this phase I clinical study was to evaluate the safety and tolerability of AWT020 monotherapy and combination with other antitumor therapies in patients with advanced malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female subjects who are at least 18 years old at the time of signing the consent form;
2. Inclusion of patients with advanced malignancies confirmed histologically or cytologically and meeting the following requirements:

   * Single-agent dose escalation and expansion phase to include patients with advanced malignant tumors who have failed or are intolerant of standard treatment, or have no standard treatment options;
   * Therapeutic effect expansion stage of single drug:

     1. NSCLC: histologically or cytologically confirmed, unresectable locally advanced, relapsed, or distant metastatic NSCLC that has progressed after prior treatment with PD-(L)1 antibody and platinum-containing chemotherapy (except after the last dose > Progression of adjuvant and neoadjuvant therapy within 6 months). Subjects with EGFR or ALK mutations will need to progress with prior treatment with appropriate kinase inhibitors.
     2. Melanoma: histologically unresectable stage III or IV melanoma that has progressed after prior chemotherapy and treatment with PD-(L)1 inhibitors (except after the last dose > Adjuvant and neoadjuvant therapy that progresses within 6 months); Mucosal melanoma does not require prior PD-(L)1 inhibitor therapy.
     3. CRC: colorectal adenocarcinoma or rectal adenocarcinoma with histologically confirmed PD-L1 composite positive score [CPS] ≥1, failure or intolerance of standard treatment, or no standard treatment options. PD-L1 expression levels in tumor tissues are based on the results of the central laboratory tests designated by the sponsor (the inclusion criteria for PD-L1 expression levels can also be adjusted according to previous data during the study).
     4. RCC: Histologically confirmed metastatic or unresectable clear cell type of RCC with disease progression after previous treatment with targeted anti-angiogenesis therapy and PD-(L)1 inhibitors.
     5. Other advanced malignancies: patients with advanced malignancies who have failed or been intolerant to standard treatment or have no standard treatment options.
   * Combination phase:

     1. NSCLC: histologically or cytologically confirmed, unresectable locally advanced, relapsed, or distant metastatic NSCLC that has not progressed after prior treatment with PD-(L)1 antibody and platinum-containing chemotherapy (except after the last dose > Progression of adjuvant and neoadjuvant therapy within 6 months). Subjects carrying EGFR or ALK mutations were allowed to progress on kinase inhibitor therapy with a previous ≤1 line.
     2. CRC: Histologically confirmed PD-L1 CPS≥1 colorectal adenocarcinoma or rectal adenocarcinoma without prior systemic therapy (except after the last dose of medication > Adjuvant therapy that progresses within 6 months); In patients with MSI-H/dMMR, previous treatment with PD-(L)1 inhibitors is permitted. PD-L1 expression levels in tumor tissues are based on the results of the central laboratory tests designated by the sponsor (the inclusion criteria for PD-L1 expression levels can also be adjusted according to previous data during the study).
     3. RCC: Histologically confirmed metastatic or unresectable clear cell RCC with disease progression after previous treatment with anti-angiogenesis targeted therapy and PD-(L)1 inhibitors.
     4. Melanoma: histologically unresectable stage III or IV melanoma that has progressed after prior chemotherapy and treatment with PD-(L)1 inhibitors (except after the last dose > Adjuvant therapy that progresses within 6 months).
     5. HCC: Histologically/cytologically confirmed or cirrhotic patients meet the clinical diagnostic criteria for HCC in AASLD, are identified as having stage B (intermediate) or stage C (advanced) BCLC HCC and are not candidates for radical surgery and/or local therapy, and have previously received PD-(L)1 inhibitors and anti-angiogenic targeted therapy progression.
     6. Other advanced malignancies: patients with advanced malignancies who have failed or been intolerant to standard treatment, or have no standard treatment options.
3. ECOG score is 0 or 1;
4. Expected survival ≥12 weeks;
5. Have at least one measurable lesion according to RECIST 1.1 evaluation criteria;
6. Good organ function;
7. Fertile female or male subjects must agree to be childfree during the study period until 6 months after the end of the last dose and voluntarily take highly effective contraception with their partner; The serum pregnancy test for WOCBP must be negative within 7 days prior to the first dose and must be non-lactation (specific contraceptive methods and WOCBP definitions are set out in section 10.3);
8. Patients participate voluntarily, give full informed consent, sign written informed consent, and have good compliance.

Exclusion Criteria:

1. Received the following drugs or treatments before the first dose:

   1. received chemotherapy, immunotherapy and other anti-tumor therapy or other investigational drugs within 21 days before the first dose, or received oral fluorouracil, small molecule targeted drugs or Chinese medicines with anti-tumor indications within 14 days before the first dose;
   2. Major surgery or radiotherapy within 28 days before the first dose (palliative radiotherapy for local bone/brain lesions allowed within 14 days before the first dose), coarse needle puncture biopsy or other minor surgery within 7 days before the start of study therapy, excluding placement of vascular infusion devices;
   3. In combination therapy, patients who have been systematically treated with corticosteroids (> 10 mg prednisone per day or equivalent) or other immunosuppressants for more than 1 week within 2 weeks prior to initial administration are allowed to be treated with inhaled or topical steroids or ≤10 mg/ day systemic prednisone and equivalent doses of similar drugs;
2. There is active central nervous system metastasis. If the patient has received radiotherapy or surgery in the past, imaging examination within 4 weeks before the first medication indicates stable brain metastases without aggravation or new neurological symptoms, hormone therapy has been discontinued 2 weeks before the first medication, and screening is allowed; For meningeal and brainstem metastases, screening is not allowed regardless of treatment.
3. Immune-related adverse events that led to permanent discontinuation occurred during previous immunosuppressive therapy (such as anti-PD -(L)1, CTLA-4, LAG-3 inhibitors, etc.);
4. There are pleural effusion, abdominal effusion or pericardial effusion with clinical symptoms that require repeated treatment (puncture or drainage, etc.);
5. There is a history of interstitial lung disease or a history of non-infectious pneumonia treated with corticosteroids, or imaging evidence of active pneumonia during the screening period;
6. The presence of severe, unhealed or split wounds, active ulcers, or untreated fractures (other than old fractures assessed by the investigator without clinical intervention);
7. Obvious bleeding tendency or severe coagulation dysfunction;
8. Have poorly controlled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure > 100 mmHg), or have a history of hypertensive crisis or hypertensive encephalopathy;
9. The toxicity of previous antitumor therapy did not return to the level ≤ Class 1 prescribed by CTCAE v5.0 or the level specified by the inclusion/exclusion criteria, except in the following cases: The related toxicity judged by the investigator to be well controlled and does not affect the safety and compliance of patients using the investigational drugs can be screened after confirmation with the sponsor;
10. Severe infection occurred within 28 days prior to administration in the first study (CTCAE v5.0> Grade 2), such as severe pneumonia, bacteremia, infection complications that require hospitalization; Active infection requiring intravenous anti-infective therapy or fever of unknown origin > 38.5℃ occurred within 2 weeks prior to the first study administration (as determined by the investigators, subjects with fever due to tumors could be enrolled);
11. Clinically significant hemoptysis for any reason (such as blood loss reaching or exceeding 50 ml/ day, or accompanied by clinical symptoms such as dyspnea and shortness of breath) or tumor bleeding (such as significant bleeding caused by tumor, manifested as hemoptysis, hematemesis, bloody stool, etc., and the blood loss reaching 50 ml/ day or more) within 1 month before the first medication, Or accompanied by anemia, hypotension, shock and other symptoms);
12. Gastrointestinal perforation, fistula, abdominal abscess, bleeding, or definite bleeding tendency (including but not limited to: severe esophagofundus varicose veins with bleeding risk, locally active digestive ulcer lesions [may be considered in investigators' assessment of ulcer stability], persistent positive stool occult blood, etc.) within 6 months before randomization; For patients with persistent positive stool occult blood, if they are patients with colorectal cancer or gastric cancer, and the positive occult blood test is believed to be related to tumor after detailed evaluation (such as local bleeding, ulcers, etc.), gastrointestinal bleeding is stable and does not cause clinical symptoms (such as anemia, hypotension, etc.) under tumor treatment or disease control, they can be considered for inclusion;
13. Severe cardiovascular and cerebrovascular diseases, including but not limited to, History of myocardial infarction, severe/unstable angina pectoris, congestive heart failure (NYHA cardiac function rating ≥2), clinically significant supratrioventricular or ventricular arrhythmia requiring pharmacological intervention, aortic aneurysm requiring surgical repair, any arterial thromboembolism/embolism event, grade 3 or higher (CTCAE) within 6 months prior to administration v5.0) Venous thrombosis/embolism events, transient ischemic attacks, cerebrovascular accidents; Left ventricular ejection fraction (LVEF) by color Doppler ultrasound < 50%. Corrected QTc> 480ms (using the Fridericia method, if the QTc is abnormal, it can be detected three times at an interval of 2 minutes, and the average value is calculated);
14. Active autoimmune diseases requiring systemic treatment (such as corticosteroids or immunosuppressive drugs) are present within 2 years prior to initial medication, including but not limited to systemic systemic lupus erythematosus, multiple sclerosis, rheumatoid arthritis, inflammatory bowel disease, vasculitis, etc. However, only thyroid, adrenal, or hypopituitarism, type 1 diabetes that can be controlled with hormone replacement therapy, psoriasis or vitiligo that does not require systemic treatment, and childhood asthma/allergies that have resolved are eligible for screening;
15. Had suffered from another malignant tumor within 5 years before the first medication; However, local tumors that have been cured are excluded, including cervical carcinoma in situ, skin basal cell carcinoma and prostate carcinoma in situ;
16. Active tuberculosis, hepatitis B (HBsAg positive with HBV DNA higher than 1000 copies /ml or 200 IU/ml), hepatitis C (HCVAb positive with HCV RNA higher than the lower limit of detection);
17. A history of immunodeficiency, including HIV testing positive, or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
18. The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participation in the study, affect treatment compliance, or interfere with the study results, patients who are judged by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
DLT rate | Up to approximately 12 months from first patient in
  DLT rate
AE | Up to approximately 12 months from first patient in
  Safety endpoint: incidence and severity of AE, abnormal changes in clinically significant laboratory and other tests
SAE | Up to approximately 12 months from first patient in
  Safety endpoint: incidence and severity of SAE, abnormal changes in clinically significant laboratory and other tests
MTD | Up to approximately 12 months from first patient in
  Determine maximum tolerated dose
RP2D | Up to approximately 32 months from first patient in
  Recommended phase II dose (RP2D) for AWT020 monotherapy and combination therapy

SECONDARY OUTCOMES:
Drug concentrations | Up to approximately 24 months from first patient in
  Drug concentrations in individual subjects at different time points after dosing
Immunogenicity | Up to approximately 24 months from first patient in
  Incidence of anti-drug antibody (ADA) and/or neutralizing antibody (Nab), titer of ADA positive samples
ORR | Up to approximately 32 months from first patient in
  Efficacy endpoint: Objective response rate(ORR) per RECIST v1.1
DOR | Up to approximately 32 months from first patient in
  Efficacy endpoint: Duration of response (DOR) per RECISIT v1.1
DCR | Up to approximately 32 months from first patient in
  Efficacy endpoint: Disease control rate (DCR) per RECISIT v1.1
PFS | Up to approximately 32 months from first patient in
  Efficacy endpoint: Progress -free survival (PFS) per RECISIT v1.1
OS | Up to approximately 32 months from first patient in
  Efficacy endpoint: Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No